CLINICAL TRIAL: NCT00473681
Title: High Blood Pressure Care for Korean Americans
Brief Title: Intervention Study to Control High Blood Pressure for Korean American
Acronym: HBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HS013160 (AHRQ)
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Self-Help Intervention Program-High Blood Pressure

SUMMARY:
The primary objective of the proposed clinical trials is to compare the differential reduction in blood pressure in underserved hypertensive adult Korean American. The study is designed to test the effectiveness of a comprehensive self-help intervention program.

DETAILED DESCRIPTION:
CVD is the leading cause of mortality among KA. Recent statistics underscoring the high prevalence and impact of uncontrolled HBP upon this population warrant the development and implementation of effective intervention. KA experiences a great deal of social isolation, which makes it more difficult for them to make behavioral changes for health improvement. individual, family, and community behaviors are part of the HBP problem and also constitute major part of the solution. The proposed research is designed to investigate these issues in a KA population and to lay the groundwork for community-based self-help health education interventions to enhance appropriate care and BP control.

Comparison(s):This community-based self-help intervention approach offers a more culturally appropriate approach to closing the health status gap for KA. Incorporating a partnership with community leaders and health and human service care providers, this approach will utilize state-of-the-art health education strategies and a well-trained bilingual nurse from the community.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as first-generation Korean American
* Age 40 to 65 years of age
* SBP≥140 or DBP≥90mmHg on HBP medication
* resident of Greater Baltimore census tracts
* Written consent to participate in the screening/eligibility visit
* SBP≥140 or DBP≥90mmHg at the KRC HBP verification visit
* Written consent to participate in the clinical trial:agreeing to participate in study data collection procedures, receiving HBP education, using HBPMT, and permitting contact with their own medical care provider.

Exclusion Criteria:

* Acute and/or terminal condition precluding participation such as terminal cancer or acute myocardial infarction
* Psychiatric diagnosis precluding participation such as schizophrenia and cognitive impairment measured by self-report, chart review, or clinical assessment.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2003-09; Primary Completion 2006-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Blood Pressure, Health-Related Quality of Life(Medical outcome Study Short Form-36) | Baseling, 12month, 24month

SECONDARY OUTCOMES:
Self-Care Behaviors of HBP Control(Hill-Bone adherence of HBP therapy scale) Enabling Skills(problem-solving skills, cognitive reframing, belief-in-self) Self-Help(Inventory of Adult Role Behaviors) | Baseline, 3months, 9 months,15 months

CONTACTS AND LOCATIONS:
Overall Officials: Miyong D Kim, PhD, Principal Investigator — Johns Hopkins university, School of Nursing
Locations (1):
- Korean Resource Center, Ellicott City, Maryland, United States

REFERENCES:
- [Background] Han HR, Kang J, Kim KB, Ryu JP, Kim MT. Barriers to and strategies for recruiting Korean Americans for community-partnered health promotion research. J Immigr Minor Health. 2007 Apr;9(2):137-46. doi: 10.1007/s10903-006-9022-x. PMID 17186370
- [Result] Kim MT, Kim EY, Han HR, Jeong S, Lee JE, Park HJ, Kim KB, Hill MN. Mail education is as effective as in-class education in hypertensive Korean patients. J Clin Hypertens (Greenwich). 2008 Mar;10(3):176-84. doi: 10.1111/j.1751-7176.2008.07571.x. PMID 18326962
- [Result] Han HR, Kim KB, Kang J, Jeong S, Kim EY, Kim MT. Knowledge, beliefs, and behaviors about hypertension control among middle-aged Korean Americans with hypertension. J Community Health. 2007 Oct;32(5):324-42. doi: 10.1007/s10900-007-9051-y. PMID 17922204
- [Result] Kim EY, Han HR, Jeong S, Kim KB, Park H, Kang E, Shin HS, Kim MT. Does knowledge matter?: intentional medication nonadherence among middle-aged Korean Americans with high blood pressure. J Cardiovasc Nurs. 2007 Sep-Oct;22(5):397-404. doi: 10.1097/01.JCN.0000287038.23186.bd. PMID 17724422
- [Derived] Han HR, Chan K, Song H, Nguyen T, Lee JE, Kim MT. Development and evaluation of a hypertension knowledge test for Korean hypertensive patients. J Clin Hypertens (Greenwich). 2011 Oct;13(10):750-7. doi: 10.1111/j.1751-7176.2011.00497.x. Epub 2011 Jul 14. PMID 21974763
- [Derived] Kim MT, Han HR, Hedlin H, Kim J, Song HJ, Kim KB, Hill MN. Teletransmitted monitoring of blood pressure and bilingual nurse counseling-sustained improvements in blood pressure control during 12 months in hypertensive Korean Americans. J Clin Hypertens (Greenwich). 2011 Aug;13(8):605-12. doi: 10.1111/j.1751-7176.2011.00479.x. Epub 2011 Jun 27. PMID 21806771
- [Derived] Kim J, Han HR, Song H, Lee J, Kim KB, Kim MT. Compliance with home blood pressure monitoring among middle-aged Korean Americans with hypertension. J Clin Hypertens (Greenwich). 2010 Apr;12(4):253-60. doi: 10.1111/j.1751-7176.2009.00218.x. PMID 20433546
- [Derived] Han HR, Kim J, Kim KB, Jeong S, Levine D, Li C, Song H, Kim MT. Implementation and success of nurse telephone counseling in linguistically isolated Korean American patients with high blood pressure. Patient Educ Couns. 2010 Jul;80(1):130-4. doi: 10.1016/j.pec.2009.10.012. Epub 2009 Nov 30. PMID 19945816